CLINICAL TRIAL: NCT04405479
Title: Spectral Analyses of Resting Postural Tremor Measured by Accelerometer and Gyroscope as a Predictive Tool of Multiple Sclerosis
Brief Title: Resting Postural Tremor in Multiple Sclerosis
Status: Recruiting | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Kamila Řasová, associate professor PhDr. Kamila Řasová, Ph.D., Charles University, Czech Republic
Other Study IDs: EK-VP/23/0/2014
Record Dates: First submitted 2020-05-20; First posted 2020-05-28 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Multiple Sclerosis
Keywords: Tremor; Accelerometer
MeSH Terms: conditions — Multiple Sclerosis; Tremor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with multiple sclerosis: MS patients will be chosen by an independent neurologist.
  Interventions: Behavioral: Examination of tremor and upper hand functions
- Healthy volunteers: Healthy controls will be paired by age and sex with MS patients.
  Interventions: Behavioral: Examination of tremor and upper hand functions

INTERVENTIONS:
Behavioral: Examination of tremor and upper hand functions — Participants will be only examined. They will not undergo any intervention.

SUMMARY:
Early diagnosis is a key factor for effective treatment of multiple sclerosis. Accelerometer and gyroscope measurement of tremor could screen potential motor control dysfunction and predict a risk for development of multiple sclerosis.

DETAILED DESCRIPTION:
The aim of this study is to test whether specially developed accelerometer and gyroscope can differentiate pattern of resting postural tremor in healthy and people with multiple sclerosis.

Spectral analysis and the correlation of the average signal spectra will be computed. Moreover, categorization based on the tremor component according to the maximum likelihood estimation will be done.

ELIGIBILITY:
Inclusion Criteria:

Group 1:

* Definite diagnosis of MS
* prevailed motor deficit of upper extremities, but without visible tremor
* stable clinical status in the preceding 3 months
* Expanded Disability Status Scale score (EDSS) ≥ 2 ≤ 7.5, and
* no corticosteroid therapy in the preceding month

Group 2:

* Healthy volunteers in the age of 20-70 years will be employed
* There will be defined as persons without any neurological disease diagnose at the time of the measurement.

Exclusion Criteria (both groups):

Patients with factors disturbing mobility (e.g. stroke, pregnancy, fractures) were excluded from the study.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People with MS and healthy volunteers
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-10-28 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Tremor | baseline
  accelerometer (1 m·s-2)

SECONDARY OUTCOMES:
Hand grip strength | baseline
  Hand dynamometer JAMA
Hand and arm function | baseline
  Nine Hole Peg Test
Psychomotor processing speed | baseline
  Coin Rotation Task

CONTACTS AND LOCATIONS:
Overall Officials: Kamila Řasová, Ph.D., Principal Investigator — Third Faculty of Mecicine, Charles Univerzity
Locations (3):
- Czechia (3):
  - Department of neurology, Prague
  - Kamila Řasová, Prague
  - Deparment of revmatology and rehabilitation, Prague

IPD SHARING:
Plan to Share IPD: No